CLINICAL TRIAL: NCT04701970
Title: Effect of Mandibular Complete Dentures Relining on Occlusal Force Distribution Using T- Scan System (A Cross-over Clinical Study)
Brief Title: Effect of Mandibular Complete Dentures Relining on Occlusal Force Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Eman Mostafa Ahmed Ibraheem, associate professor, National Research Centre, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11010203
Record Dates: First submitted 2020-11-23; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Occlusion
Keywords: complete dentures; relining; occlusal force; T scan system
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: occlusal load distribution was measured by T scan system before and after mandibular complete denture relining with soft denture liner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- changes in the occlusal load distribution (Other): A crossover clinical study was carried out with previously constructed and used conventional complete dentures before relining with soft denture liners and then with the same dentures after relining with soft denture liners. patients were comfortably using their relined mandibular complete dentures for at least three months and the retention and stability of the conventional dentures were assessed before second recording of occlusal parameter. The evaluation of occlusal force distribution was carried out with the aid of T-Scan device
  Interventions: Procedure: relining of mandibular complete denture

INTERVENTIONS:
Procedure: relining of mandibular complete denture — Relining of mandibular dentures was performed by reducing one mm of the denture fitting surfaces and borders to make a right-angled border. apply two separate layers of Mucopren adhesive upon the vestibular surface of the mandibular denture and allow each layer to dry for about 40 seconds. then, the lower denture was inserted and molded in patient mouths; while biting in centric occlusion with the opposing maxillary complete dentures.

SUMMARY:
evaluation of occlusal force distribution was carried out with the aid of T-Scan device (Tekscan Inc., South Boston, MA, USA) for mandibular complete dentures before and after relining with long term soft liner for controlled type 2 diabetic patients.

DETAILED DESCRIPTION:
A crossover clinical study was carried out with previously constructed and used conventional complete dentures before relining with soft denture liners and then with the same dentures after relining with soft denture liners. The study sample included 50 males completely edentulous contributors, All patients were controlled type 2 diabetes during the study period. All selected patients had previously constructed and used conventional heat cured acrylic resin complete dentures for not less than two years with history of retention and stability problems of mandibular dentures. Mandibular complete dentures had received the essential prosthetic adjustments aiming to achieve optimal retention, maximum stability and the necessary occlusal contacts. The first occlusal parameters were recorded before denture relining. Relining of mandibular dentures was performed and Patients were comfortably using their relined mandibular complete dentures for at least three months and the retention and stability of the conventional dentures were assessed before second recording of occlusal parameter. The evaluation of occlusal force distribution was carried out with the aid of T-Scan device (Tekscan Inc., South Boston, MA, USA). The first record was recorded before denture relining and the second record was three months after denture relining

ELIGIBILITY:
Inclusion Criteria:

* All patients were controlled type 2 diabetes
* All patients were non-smokers
* had an Angle class I maxillo-mandibular relationship.
* Patients having moderately developed maxillary and mandibular alveolar ridges lined with firm mucoperiostea.

Exclusion Criteria:

* history of temporomandibular disorders, or neuromuscular disorders like; bruxism or severe clenching
* presence of medical problems or severe chronic diseases
* any intraoral soft or hard tissue pathology.

Ages: 49 Years to 63 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
assessment of the effect of relining of mandibular complete dentures with soft relining material on occlusal force distribution using T-Scan system. load distribution for 50 completely edentulous patient before and after complete denture relining | for each participant: the complete denture should be worn for three months
  Fifty completey edentulous patients having previously constructed and utilized conventional complete dentures were selected for this study. Relining of mandibular complete dentures with soft denture liner was carried out. Distribution of occlusal force was evaluated with the aid of T-Scan device before denture relining and three months after relining.
  measured before relining of complete denture with soft liner and measured again after complete denture relining.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, El- Dokki, Egypt